CLINICAL TRIAL: NCT06220565
Title: Evaluation of Product Effectiveness of a Graded Exercise Intervention for Patients With Knee Osteoarthritis in a Community Scenario
Brief Title: Evaluation of Product Effectiveness of the Intervention for Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhu Dian, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MDH0002
Record Dates: First submitted 2024-01-12; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee; Product Use Issue; Sports Physical Therapy
Keywords: Older adults; Osteoarthritis; Sports Rehabilitation; Product Design
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Products for graded exercise interventions "Graded Exercise" (Experimental): Through digital means, patients are able to execute a personalized exercise program based on their rehabilitation plan and incorporate digital assessment methods to receive real-time feedback and recommendations for adjustments. By providing a personalized rehabilitation program and regular telecare, the aim is to focus on the patient's rehabilitation needs in a holistic manner.
  Interventions: Device: sensor and wearable device "Graded Exercise"; Other: exercise
- Education group (Placebo Comparator): Educational Manual on Exercise Rehabilitation for Patients with Osteoarthritis of the Knee
  Interventions: Other: exercise; Other: Educational Manual

INTERVENTIONS:
Device: sensor and wearable device "Graded Exercise" — The program plans to use rational mechanism to provide safe and targeted exercise interventions to patients at different stages of their lives through three aspects: education, motivation and feedback. Through real-time collection of knee function parameters, real-time feedback on the effect of exercise intervention, and tracking the changes in the functional status of patients' knee joints. On the basis of improving knee function, we further improve patients' compliance with exercise intervention.
  Considering the community scenario, we plan to use sensors and wearable devices to realize the function of the knee joint on the basis of the existing technology. wearable devices to realize the digital assessment of knee function to reduce patient's time and cost and improve efficiency. At the same time, this digital assessment will provide a basis for decision-making for patient self-management.
  Arms: Products for graded exercise interventions "Graded Exercise"
Other: exercise — exercise
Other: Educational Manual — Educational Manual
  Arms: Education group

SUMMARY:
Osteoarthritis of the knee is a common, chronic joint pathology that causes participants to suffer from pain, dysfunction, and reduced quality of life. The goal is to improve the quality of life and rehabilitation of patients by making rehabilitation exercises electronic and the system can be personalized to their specific conditions.

The focus of this study was on exercise interventions, and an interactive software was designed that combines repetitive motion and real-time feedback mechanisms. The software provides a series of rehabilitation movements that are specific to the characteristics of osteoarthritis of the knee in older adults, aiming to help participants gradually improve joint range of motion and muscle strength through exercise. The real-time feedback mechanism, on the other hand, monitors the participants' exercise status in real time through wearable devices, providing intuitive feedback to the participants to ensure that they perform the rehabilitation movements correctly, thus ensuring the scientificity and safety of the exercise.

In this study, investigators designed an exercise assessment and exercise intervention system for patients with knee osteoarthritis. In the exercise assessment part, the study combines several tools. First, the WOMAC scale was used to systematically assess patients' joint pain, stiffness, and dyskinesia. Second, physical function tests are used to assess the patient's overall exercise capacity, including indicators such as the number of sit-ups and rises. In addition, a wearable device was designed in this paper for real-time collection of knee angle information.

ELIGIBILITY:
Inclusion Criteria:

1. Those who meet the diagnostic criteria for osteoarthritis and are diagnosed with osteoarthritis of the knee;
2. Age greater than grade 18 years old;
3. Good communication and comprehension skills, able to understand the questionnaire clearly;
4. Informed consent and willingness to participate in the study.

Exclusion Criteria:

1. Patients with knee pain caused by other diseases;
2. Patients with severe knee pain and discomfort;
3. Patients with severe organic lesions of vital organs such as heart, brain and kidney;
4. Patients who have been treated with knee replacement.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
University of Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | 10 minutes
  The WOMAC scale provides a better assessment of elderly and chronic patients. The scale consists of 3 dimensions: pain, morning stiffness, and dysfunction, with a total of 24 items, including 5 items for pain and 2 items for morning stiffness. The scale consists of 3 dimensions: pain, morning stiffness, and dysfunction, with a total of 24 items, of which 5 are for pain, 2 for morning stiffness, and 17 for dysfunction, and can be completed within 5-10 min.

SECONDARY OUTCOMES:
Affective State Depression Rating Scale for Older Adults | 10 minutes
  A total of 30 entries represent the core of geriatric depression and include the following symptoms: low mood, decreased activity, irritability, withdrawal from painful thoughts, negative evaluations of the past, present, and future. Negative evaluations of the past, present and future.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Zhao, Dr, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Dian Zhu, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu T, Han T, Zhu D. Effects of Resistance Exercise Combined with Cognitive Intervention Therapy on Cognitive Decline: A Randomized Controlled Trial of a Cognitively Declining Elderly Population. Games Health J. 2025 Aug;14(4):281-294. doi: 10.1089/g4h.2024.0055. Epub 2024 Nov 27. PMID 39605293